CLINICAL TRIAL: NCT00224289
Title: Effect of Age on Efficacy and Response Time of Latanoprost 0.005% in Patients With Glaucoma
Brief Title: Effect of Age on Latanoprost 0.005% in Patients With Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27390
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-11

CONDITIONS: Glaucoma
Keywords: Latanoprost; Glaucoma; Intraocular pressure
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): All participants will be taking Latanoprost; This study compares efficacy within age groups.
  Interventions: Drug: Latanoprost 0.005%

INTERVENTIONS:
Drug: Latanoprost 0.005% — Latanoprost 0.005% ophthalmic solution QHS 8 weeks
  Other Names: Xalatan

SUMMARY:
Latanoprost is a commonly used treatment for glaucoma. Because of its mechanism of action, it is plausible that the age of a patient using the medication may affect its efficacy and time of onset.

We are going to study the effectiveness of Latanoprost in people of different ages, to see if it changes based on the age of the patient.

DETAILED DESCRIPTION:
Latanoprost is a topical ocular hypotensive medication with a well established safety and efficacy profile. Its effect is mediated by an increase in uveoscleral outflow, due to enzymatic degradation of the extracellular matrix within the ciliary muscle. Since the amount of extracellular matrix within the human eye increases with age, and uveoscleral outflow decreases with age, it would be expected that there should be a difference in the efficacy of latanoprost in patients of different ages. This has not been demonstrated in studies assessing the overall effect of latanoprost across adult age groups using multivariate analysis. (Camras CB et al, 1996).

However, a difference in timing of onset of drug effect may get overlooked in clinical studies and in clinical practice as well, as patients tend to be seen from two to eight weeks after initiation of treatment, by which time any differences in response time may have already occurred and leveled off.

To our knowledge, there are no studies specifically looking at the timing of onset of drug effect of latanoprost in different age groups. Because of the theoretical plausibility of this effect based on the mechanism of action of latanoprost, this represents an opportunity to further elucidate the characteristics of this medication in a manner which has clinical and scientific relevance.

Our aim is thus to determine if there is a difference in timing of onset of the ocular hypotensive effect of latanoprost in glaucoma patients of different age groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of open angle glaucoma,
* pseudoexfoliation glaucoma, pigmentary glaucoma or ocular hypertension in one or both eyes;
* IOP above their target pressure as determined by a glaucoma specialist;
* willingness to participate in the study.

Exclusion Criteria:

* hypersensitivity to any of the components of the treatment medication;
* previous use of topical prostaglandins;
* documented ocular infection or intraocular inflammation within the past year;
* previous filtering surgery or complicated cataract surgery;
* active corneal disease;
* presence of cystoid macular edema;
* laser trabeculoplasty or any other ocular laser procedure within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shields, MD, Principal Investigator — Yale University
Locations (1):
- Yale Eye Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Latanoprost: All participants will be taking Latanoprost; This study compares efficacy within age groups.
  Latanoprost 0.005% : Latanoprost 0.005% ophthalmic solution QHS 8 weeks
Period: Overall Study
Arm/Group | Topical Latanoprost
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Topical Latanoprost
Number analyzed (Participants) | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 61.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Pre-Treatment IOP (Intraocular Pressure)
Description: Subjects applied topical latanoprost at bedtime for 8 weeks
Time Frame: At baseline (before treatment)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Topical Latanoprost
Number analyzed (Participants) | 17
mm Hg | 21.8 (6.28)

2. Primary Outcome: Post-Treatment IOP (Intraocular Pressure)
Description: Subjects applied topical latanoprost at bedtime for 8 weeks
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Topical Latanoprost
Number analyzed (Participants) | 17
mm Hg | 18.3 (5.36)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected for 8 weeks per subject. The subjects received the study medication for 8 weeks.
Arm/Group | Topical Latanoprost
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topical Latanoprost (N=17)
Red Eye w/ Foreign Body Sensation (Eye disorders) | 1
Eye Tearing (Eye disorders) | 1
Blurry Vision (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes